CLINICAL TRIAL: NCT02766504
Title: Ultrasound in Airway Assessment of Morbidly Obese Patients
Acronym: AiUs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Other Study IDs: refa 7 105
Record Dates: First submitted 2015-10-03; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: General Anesthesia of Morbid Obese Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: airway ultrasound — airway assessment using ultrasound

SUMMARY:
the study aims to evaluate the role of airway ultrasound as a new evolving modality in assessment and management of airway in surgical patients

ELIGIBILITY:
Inclusion Criteria:

* all surgical list patients planned for general anesthesia from october 2015 to may 2016

Exclusion Criteria:

* Patient refusal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: surgical list patients with indicated endotracheal tube insertion for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
prediction of difficult intubation in morbid obese patients | during endotracheal tube insertion
  prediction of difficult intubation in morbid obese versus traditional airway scores; Mallampati score.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt